CLINICAL TRIAL: NCT01542268
Title: Effect of Pentoxifylline on Tight Junctions of Intestinal Mucosa in Patients With Irritable Bowel Syndrome
Brief Title: Effect of Pentoxifylline on Tight Junctions (TJs) of Intestinal Mucosa in Patients With Irritable Bowel Syndrome(IBS)
Acronym: IBS-PTX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBS-PTX
Record Dates: First submitted 2011-09-23; First posted 2012-03-02 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: pentoxifylline; tight junction signalling; intestinal epithelial barrier; irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pentoxifylline (Active Comparator)
  Interventions: Drug: pentoxifylline
- pentoxifylline placebo (Placebo Comparator)
  Interventions: Drug: pentoxifylline placebo

INTERVENTIONS:
Drug: pentoxifylline — Patients will take 800mg/day, via oral, of pentoxifylline. 400 mg of pentoxifylline each 12 hours (during meals time).Period: 3 months.
  Other Names: A
  Arms: pentoxifylline
Drug: pentoxifylline placebo — Patients will take 800mg/day, via oral, of pentoxifylline placebo. 400 mg of pentoxifylline placebo each 12 hours (during meals time).Period: 3 months.
  Other Names: B
  Arms: pentoxifylline placebo

SUMMARY:
The purpose of this study is to determine the therapeutics effectiveness of oral pentoxifylline treatment in patients with IBS.

DETAILED DESCRIPTION:
Disruption of the intestinal epithelial barrier is part of the pathophysiology of IBS favoring immune activation present in the mucosa of these patients and the development of symptoms in IBS. To evaluate the effect of treatment with pentoxifylline (PTX) in patients with IBS related to clinical response and modulation of the components of the epithelial barrier at the level of intestinal mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* Most of the patient with IBS will be chose between the patients who go to Digestive System ambulatory external medical office from our Center.
* Be studied and with clinical monitoring al least 6 months before be included.
* Fulfill with Roma III Criteria for IBS (Gastroenterology 2006;130:1377-90) with moderate-severe seriousness according to Modification Francis Scale

Exclusion Criteria:

* 2 weeks before colon biopsia, any patient cann´t take salicylates, NSAID, antibiotics,anticholinergics,opiates or any other medication / product for asintomatic treatment of diarrea.
* 3 months before colon biopsia, any patient cann´t take medicaments as corticoides, antihistamines or immunosuppressive
* 6 months before colon biopsia, any patient cann´t recive radiotherapy or chemotherapy.
* Pentoxifilina Alergic Reactions
* Pregnants
* Grave kidney failure
* Grave Hepatic failure
* Menthal or legal disability to sign the consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Severity of abdominal pain | 3 months from the first day of treatment
  Clinical endpoint:
  Average daily severity of abdominal pain on a 0-10 scale [ Time Frame: Week 0 to week 12 ] [ Designated as safety issue: No ] Days with urgency [ Time Frame: Week 0 to week 12 ] [ Designated as safety issue: No ] Mean stool consistency using Bristol Stool Form Score [ Time Frame: Week 0 to week 12 ] [ Designated as safety issue: No ] Global satisfaction with control of IBS symptoms as assessed from the answer to the question "Have you had satisfactory relief of your IBS symptoms this week? Yes / No. "

SECONDARY OUTCOMES:
Mucosal byopsies | 3 months from the first day of treatment
  Effect of pentoxifylline treatment from mucosal byopsies on:
  1. epithelial morphology;
  2. mucosal immune cell subsets;
  3. changes of gene expression of genes related to intestinal epithelial barrier component( tight junctions)

CONTACTS AND LOCATIONS:
Overall Officials: LAURA RAMOS, MD, Principal Investigator — COMPLEJO HOSPITALARIO UNIVERSITARIO DE CANARIAS
Locations (1):
- Complejo Hospitalario Universitario de Canarias, San Cristóbal de La Laguna, S/c Tenerife, Spain